CLINICAL TRIAL: NCT02160587
Title: A Clinical Evaluation of the Contact Sensitizing Potential of Topically Applied ZuraPrep™ and ZuraPrep™ Without IPA in Healthy Adult Volunteers
Brief Title: Safety Study to Evaluate the Contact Sensitizing Potential of Topically Applied ZuraPrep™ and ZuraPrep™ Without IPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zurex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: 130821-303 (ZX-ZP-0018)
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — chlorhexidine gluconate; citrate, isopropyl alcohol, methylene blue, parabens drug combination; 2-Propanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZuraPrep (Active Comparator): Irritation scores of the following applied to test sites will be compared: ZuraPrep, ZuraPrep without IPA, ChloraPrep, and 0.9% Physiological Saline.
  Interventions: Drug: Chloraprep; Drug: 0.9% Physiological Saline; Other: ZuraPrep without IPA

INTERVENTIONS:
Drug: Chloraprep — ChloraPrep will be compared to ZuraPrep with regard to skin sensitization and irritation.
  Other Names: Reference Product; 2% Chlorhexidine Gluconate and 70% IPA
Drug: 0.9% Physiological Saline — 0.9% Physiological Saline will be compared to ZuraPrep with regard to skin sensitization and irritation.
  Other Names: Negative Control
Other: ZuraPrep without IPA — ZuraPrep without IPA will be compared to ZuraPrep with regard to skin sensitization and irritation
  Other Names: ZuraPrep without Isopropyl Alcohol (IPA)

SUMMARY:
This is a safety study to determine the skin sensitization potential of ZuraPrep™ and ZuraPrep™ without isopropyl alcohol (IPA) after repetitive patch applications to skin of human subjects. Indications of both sensitization and skin irritation will be evaluated.

DETAILED DESCRIPTION:
This study is designed to determine if the test product, ZuraPrep™ is a skin sensitizing agent when applied to human skin. The study, a modified Draize skin sensitization evaluation, will be conducted in three discrete phases: 1) induction, 2) rest, and 3) challenge. During the Induction Phase, skin sites are exposed to the test product repeatedly for 21 consecutive days. The Rest Phase, a 14-day period when no treatment is performed, serves to provide adequate time for the immune system to react to ZuraPrep™, given any of its components serve as antigens. During the Challenge Phase, the subjects' skin is re-exposed to the test product (ZuraPrep™) to determine if it is likely to be immunosensitizing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, at least 18 years of age and of any race
* Subjects must be free of tattoos, sunburn, dermatoses, cuts, lesions or other disorders of the skin of the back.
* Subjects must be in good general health

Exclusion Criteria:

* Known allergies to latex, metals, tape and/or adhesives, soap, citric acid, methylene blue, methylparaben, propylparaben, chlorhexidine gluconate, isopropyl alcohol, and sodium lauryl sulfate.
* Exposure of the back region to antimicrobial agents, medicated soaps, medicated shampoos, medicated lotions, strong detergents, sun-tanning, use of tanning beds, or swimming or soaking in pools or hot tubs, in the 7 days prior to, or during the 3-week test period.
* Use of topical or systemic corticosteroid, antihistamine, or anti-inflammatory medications in the 7 days prior to, or during the 3-week test period.
* Current or recent severe illness such as asthma, diabetes, hepatitis, organ transplant, mitral valve prolapse, congenital heart disease, internal prostheses, or any immunocompromised condition such as AIDS or HIV positive.
* Pregnancy, plans to become pregnant, breast-feeding
* Any active skin rash or breaks in the skin of the back
* Any sunburn or tattoos on the skin of the back
* Current active skin disease or inflammatory skin condition including contact dermatitis
* Participation in a clinical study in the past 7 days or current participation in another clinical study
* Any medical condition or use of any medications that, in the opinion of the Principal Investigator, would preclude participation
* Unwillingness to fulfill the performance requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Skin sites evaluated and graded for irritancy or sensitization | 0-40 days post dose
  Only frank sensitization will be categorized, as a positive control (known sensitizing agent) is prohibitive due to ethical considerations/risk of life-time sensitization. Reactions observed will be assessed as to whether indicative of sensitization or of irritation.

SECONDARY OUTCOMES:
Statistics of irritation scores | 0-40 days post dose
  Irritation scores, relative to the Test Products, Reference Product, and the Negative Control applied to skin on each test day will be compared as well as the total cumulative irritation scores across all test days.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Butler, PhD, Principal Investigator — BioScience Laboratories, Inc.
Locations (1):
- BioScience Laboratories, Inc., Bozeman, Montana, United States